CLINICAL TRIAL: NCT00700102
Title: A Randomized, Open-label Phase III Intergroup Study: Effect of Adding Bevacizumab to Cross Over Fluoropyrimidine Based Chemotherapy (CTx) in Patients With Metastatic Colorectal Cancer and Disease Progression Under First-line Standard CTx/Bevacizumab Combination
Brief Title: A Study of Avastin (Bevacizumab) Plus Crossover Fluoropyrimidine-Based Chemotherapy in Patients With Metastatic Colorectal Cancer.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML18147; 2006-004634-32 (EudraCT Number)
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2015-07-30 (Estimated); Last update posted 2015-07-30 (Estimated); Status verified 2015-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Drug Therapy; Bevacizumab

ARMS (2):
- Chemotherapy (Active Comparator): Chemotherapy alone until disease progression, unacceptable toxicity, or patient refusal
  Interventions: Drug: Chemotherapy
- Chemotherapy + Bevacizumab (Experimental): Chemotherapy and Bevacizumab until disease progression, unacceptable toxicity, or patient refusal
  Interventions: Drug: Chemotherapy; Drug: Bevacizumab

INTERVENTIONS:
Drug: Chemotherapy — As prescribed
Drug: Bevacizumab — Bevacizumab, 5 mg/kg intravenously (IV) on days 1 and 14 of each 4 week cycle, or 7.5 mg/kg IV on days 1 and 22 of each 6 week cycle.
  Other Names: Avastin
  Arms: Chemotherapy + Bevacizumab

SUMMARY:
This study will evaluate the efficacy and safety of adding bevacizumab to crossover fluoropyrimidine-based chemotherapy in patients with metastatic colorectal cancer who have experienced disease progression under first line treatment with standard chemotherapy plus bevacizumab. Participants will receive chemotherapy alone, or in combination with bevacizumab. The anticipated time on study treatment is until disease progression or unacceptable toxicity occurs. Participants are allowed to continue on bevacizumab, even after stopping chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=18 years of age
* Metastatic colorectal cancer and disease progression
* Previously treated with first-line chemotherapy plus Avastin
* Eastern Cooperative Oncology Group (ECOG) performance status <=2.

Exclusion Criteria:

* Diagnosis of progression of disease more than 3 months after last Avastin administration
* First-line patients with progression-free survival in first-line of <3 months
* Patients receiving less than 3 consecutive months of Avastin in first-line therapy
* Past or current history (within the last 2 years prior to treatment start) of other malignancies, except for curatively treated basal and squamous cell cancer of the skin or in situ cancer of the cervix
* Clinically significant cardiovascular disease within 6 months prior to start of study treatment
* Known central nervous system (CNS) disease, except for treated CNS metastases as defined by protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2006-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (248):
- Austria (19):
  - Dornbirn
  - Fürstenfeld
  - Graz
  - Hall in Tirol
  - Innsbruck
  - Krems
  - Leoben
  - Linz
  - Rankweil
  - Ried-innkreis
  - Salzburg
  - Sankt Pölten
  - Sankt Veit an der Glan
  - Steyr
  - Vienna
  - Villach
  - Waidhofen A D Thaya
  - Wels
  - Wiener Neustadt
- Belgium (6):
  - Aalst
  - Assebroek
  - La Louvière
  - Leuven
  - Liège
  - Turnhout
- Czechia (3):
  - Brno
  - Olomouc
  - Prague
- Denmark (6):
  - Copenhagen
  - Esbjerg
  - Herlev
  - Herning
  - Hillerød
  - Næstved
- Estonia (2):
  - Tallinn
  - Tartu
- Finland (5):
  - Helsinki
  - Oulu
  - Tampere
  - Turku
  - Vaasa
- France (66):
  - Agen
  - Albi
  - Amiens
  - Amilly
  - Antibes
  - Antony
  - Arras
  - Avignon
  - Besançon
  - Béziers
  - Bordeaux
  - Bourgoin
  - Caen
  - Cahors
  - Chambray-lès-Tours
  - Clermont-Ferrand
  - Colmar
  - Compiègne
  - Dechy
  - Dijon
  - Grenoble
  - La Roche-sur-Yon
  - La Seyne-sur-Mer
  - Lagny-sur-Marne
  - Le Kremlin-Bicêtre
  - Le Mans
  - Libourne
  - Lille
  - Limoges
  - Lliie
  - Longjumeau
  - Lyon
  - Marseille
  - Mâcon
  - Meaux
  - Metz
  - Mont-de-Marsan
  - Montbéliard
  - Montfermeil
  - Montpellier
  - Mougins
  - Nancy
  - Nantes
  - Neuilly-sur-Seine
  - Nevers
  - Nice
  - Orléans
  - Paris
  - Pessac
  - Périgueux
  - Pierre-Bénite
  - Pontoise
  - Reims
  - Rennes
  - Rodez
  - Rouen
  - Saint-Brieuc
  - Saint-Cloud
  - Saint-Grégoire
  - Saint-Herblain
  - Saint-Nazaire
  - Senlis
  - Strasbourg
  - Suresnes
  - Vandœuvre-lès-Nancy
  - Verdun
- Germany (83):
  - Aachen
  - Aschaffenburg
  - Augsburg
  - Bergisch Gladbach
  - Berlin
  - Bietigheim
  - Bochum
  - Bonn
  - Bremen
  - Chemnitz
  - Cologne
  - Darmstadt
  - Dessau
  - Dortmund
  - Dresden
  - Duisburg
  - Erlangen
  - Eschweiler
  - Essen
  - Esslingen am Neckar
  - Flensburg
  - Frankfurt
  - Frechen
  - Fulda
  - Geilenkirchen
  - Gifhorn
  - Greifswald
  - Gummersbach
  - Halle
  - Hamburg
  - Hanover
  - Heidelberg
  - Heidenheim
  - Hildesheim
  - Hof
  - Homburg/Saar
  - Kassel
  - Köthen
  - Kronach
  - Laatzen
  - Leer
  - Lehrte
  - Leipzig
  - Lemgo
  - Leverkusen
  - Limburg
  - Ludwigsburg
  - Lübeck
  - Magdeburg
  - Magedburg
  - Mainz
  - Mannheim
  - Marburg
  - Marktredwitz
  - Marl
  - Moers
  - Mönchengladbach
  - Mutlangen
  - Mülheim
  - München
  - Münster
  - Neunkirchen/Saar
  - Neustadt
  - Nordhausen
  - Oldenburg
  - Olpe
  - Pinneberg
  - Regensburg
  - Remscheid
  - Rostock
  - Rotenburg (Wümme)
  - Rötha
  - Schönebeck
  - Schwerin
  - Stade
  - Stuttgart
  - Suhl
  - Troisdorf
  - Ulm
  - Velbert
  - Wernigerode
  - Wiesbaden
  - Würselen
- Netherlands (4):
  - Amersfoort
  - Capelle aan den IJssel
  - Leiden
  - Tilburg
- Norway (5):
  - Ålesund
  - Bergen
  - Kristiansand
  - Lorenskog
  - Oslo
- Portugal (4):
  - Aveiro
  - Coimbra
  - Lisbon
  - Porto
- Saudi Arabia (3):
  - Dammam
  - Jeddah
  - Riyadh
- Spain (32):
  - Alicante, Alicante
  - Elche, Alicante
  - Elda, Alicante
  - Torrevieja, Alicante
  - Palma de Mallorca, Balearic Islands
  - Barcelona, Barcelona
  - Manresa, Barcelona
  - Sabadell, Barcelona
  - Sant Cugat del Vallès, Barcelona
  - Burgos, Burgos
  - Cadiz, Cadiz
  - Santander, Cantabria
  - Castellon, Castellon
  - Córdoba, Cordoba
  - Girona, Girona
  - Granada, Granada
  - Donostia / San Sebastian, Guipuzcoa
  - Huelva, Huelva
  - A Coruña, La Coruña
  - Lleida, Lerida
  - Alcorcón, Madrid
  - Madrid, Madrid
  - Parla, Madrid
  - Murcia, Murcia
  - Navarra, Navarre
  - Oviedo, Principality of Asturias
  - Seville, Sevilla
  - Reus, Tarragona
  - Sagunto, Valencia
  - Valencia, Valencia
  - Bilbao, Vizcaya
  - Zaragoza, Zaragoza
- Sweden (3):
  - Lund
  - Uppsala
  - Vaxjo
- Switzerland (7):
  - Aarau
  - Basel
  - Bern
  - Chur
  - Lucerne
  - Winterthur
  - Zurich

REFERENCES:
- [Derived] Li Y, Hu M, Zhang Z, Chu M, Xu R, Liu L, Dong W, Yang M, Zhang R. Cost-effectiveness analysis of continuing bevacizumab plus chemotherapy versus chemotherapy alone after first progression of metastatic colorectal cancer. Cancer Med. 2024 Jan;13(1):e6904. doi: 10.1002/cam4.6904. Epub 2024 Jan 8. PMID 38186268
- [Derived] Kubicka S, Greil R, Andre T, Bennouna J, Sastre J, Van Cutsem E, von Moos R, Osterlund P, Reyes-Rivera I, Muller T, Makrutzki M, Arnold D; ML18147 study investigators including AIO, GERCOR, FFCD, UNICANCER GI, TTD, BGDO, GEMCAD, and AGMT groups. Bevacizumab plus chemotherapy continued beyond first progression in patients with metastatic colorectal cancer previously treated with bevacizumab plus chemotherapy: ML18147 study KRAS subgroup findings. Ann Oncol. 2013 Sep;24(9):2342-9. doi: 10.1093/annonc/mdt231. Epub 2013 Jul 12. PMID 23852309
- [Derived] Bennouna J, Sastre J, Arnold D, Osterlund P, Greil R, Van Cutsem E, von Moos R, Vieitez JM, Bouche O, Borg C, Steffens CC, Alonso-Orduna V, Schlichting C, Reyes-Rivera I, Bendahmane B, Andre T, Kubicka S; ML18147 Study Investigators. Continuation of bevacizumab after first progression in metastatic colorectal cancer (ML18147): a randomised phase 3 trial. Lancet Oncol. 2013 Jan;14(1):29-37. doi: 10.1016/S1470-2045(12)70477-1. Epub 2012 Nov 16. PMID 23168366

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study enrolled 820 patients at 220 sites located in 15 countries in Europe and Saudi Arabia. Study AIO KRK 0504 enrolled 261 patients, and 559 patients subsequently enrolled in Study ML18147 when the study was transferred to Hoffmann LaRoche (in 2008).
Period: Overall Study
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Started | 411 | 409
Intention to Treat | 410 | 409
Received at Least One Dose | 407 | 403
Completed | 9 | 14
Not Completed | 402 | 395
Not completed — Died | 394 | 385
Not completed — Lost to Follow-up | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab | Total
Number analyzed (Participants) | 411 | 409 | 820
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.55) | 62.1 (9.78) | 62.0 (9.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 152 | 142 | 294
  Male | 259 | 267 | 526

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival: Time From Randomization to Death From Any Cause
Time Frame: within 6.5 years
Population: Intention to treat
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 410 | 409
months | 9.8 [9 to 11] | 11.2 [10 to 12]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.0062, Log Rank; Hazard Ratio (HR) = 0.81, 95% CI 2-sided [0.69 to 0.94]

2. Secondary Outcome: Overall Survival: Months From Time of First Line Therapy
Time Frame: within approximately 9.6 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 410 | 409
months | 22.5 [21 to 25] | 23.9 [22 to 26]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Kaplan Meier Estimate; Test type: Superiority or Other; p = 0.1713, Log Rank; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.77 to 1.05]

3. Secondary Outcome: Participants With Progression Free Survival Event
Time Frame: within 6.5 years
Population: Unstratified intention to treat population
Measure: Number; unit: participants
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 410 | 409
participants | 394 | 386

4. Secondary Outcome: Progression Free Survival: Time to Event
Time Frame: within 6.5 years
Population: Unstratified intention to treat population
Measure: Median (Full Range); unit: Months
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 410 | 409
Months | 4.1 [0 to 27] | 5.7 [0 to 38]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p < .0001, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.59 to 0.78]

5. Secondary Outcome: Response Rate: Percentage of Participants With Best Overall Response, Defined as Confirmed Complete Response (CR) or Partial Response (PR) According to RECIST Criteria
Time Frame: within 6.5 years
Population: Participants with measurable disease
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 406 | 404
percentage of participants | 3.9 [2.3 to 6.3] | 5.4 [3.4 to 8.1]
Statistical Analysis 1: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.3113, Chi-squared; Mean Difference (Final Values) = 1.50, 95% CI 2-sided [-1.5 to 4.5]
Statistical Analysis 2: Comparison: Chemotherapy vs Chemotherapy + Bevacizumab; Test type: Superiority or Other; p = 0.4315, Cochran-Mantel-Haenszel

6. Secondary Outcome: Response Rate: Participants With Response Status Based on RECIST Criteria
Description: Response Evaluation Criteria In Solid Tumors (RECIST) is a set of published rules that define when tumors in cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progress") during treatment.
Time Frame: within 6.5 years
Population: Participants with measurable disease
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Number analyzed (Participants) | 406 | 404
percentage of participants
  Complete response | 0.5 [0.1 to 1.8] | 0.2 [0.0 to 1.4]
  Partial response | 3.4 [1.9 to 5.7] | 5.2 [3.2 to 7.8]
  Stable Disease | 50.2 [45.3 to 55.2] | 62.6 [57.7 to 67.4]
  Progressive Disease | 35.0 [30.3 to 39.8] | 21.5 [17.6 to 25.9]
  Missing (No Response Assessment) | 10.8 [NA to NA] — Missing data not analyzable | 10.4 [NA to NA] — Missing data not analyzable

ADVERSE EVENTS:
Time Frame: First subject first visit to end of trial within 7.25 years
Description: Safety Analysis Set was defined as all randomized patients who received any amount of study treatment, and were analyzed according to actual treatment received.
Arm/Group | Chemotherapy | Chemotherapy + Bevacizumab
Serious Adverse Events (participants affected / at risk) | 137/409 | 130/401
Other Adverse Events (participants affected / at risk) | 379/409 | 382/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=409) | Chemotherapy + Bevacizumab (N=401)
Abdominal hernia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 9 (9) | 6 (6)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 1 (1)
Ascites (Gastrointestinal disorders) | 2 (2) | 1 (1)
Colonic obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 16 (16) | 13 (13)
Enteritis (Gastrointestinal disorders) | 0 (0) | 3 (3)
Enterovesical fistula (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (2)
Gastrointestinal hopomotility (Gastrointestinal disorders) | 0 (0) | 2 (3)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 4 (4) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Inguinal hernia, obstructive (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 2 (2)
Intestinal perforation (Gastrointestinal disorders) | 1 (1) | 4 (4)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 3 (4)
Oesophagitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Proctalgia (Gastrointestinal disorders) | 0 (0) | 1 (3)
Rectal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 4 (4) | 7 (7)
Subileus (Gastrointestinal disorders) | 2 (2) | 7 (8)
Sepsis (Infections and infestations) | 5 (6) | 2 (2)
Infection (Infections and infestations) | 3 (3) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3)
Device related infection (Infections and infestations) | 1 (1) | 3 (3)
Febrile infection (Infections and infestations) | 2 (3) | 0 (0)
Urosepsis (Infections and infestations) | 1 (1) | 2 (2)
Anal abscess (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1)
Abdominal abscess (Infections and infestations) | 1 (1) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0)
Clostridium difficile infection (Infections and infestations) | 1 (1) | 0 (0)
Device related sepsis (Infections and infestations) | 0 (0) | 1 (1)
Enterococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis clostridial (Infections and infestations) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 1 (1)
Staphylococcal sepsis (Infections and infestations) | 0 (0) | 1 (1)
Systemic candida (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 11 (13) | 7 (10)
Disease progression (General disorders) | 4 (4) | 3 (3)
General physical health deterioration (General disorders) | 1 (1) | 3 (3)
Chest pain (General disorders) | 1 (1) | 2 (2)
Fatigue (General disorders) | 2 (2) | 1 (1)
Mucosal inflammation (General disorders) | 1 (1) | 2 (2)
Asthenia (General disorders) | 2 (2) | 0 (0)
Obstruction (General disorders) | 2 (2) | 0 (0)
Device breakage (General disorders) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 1 (1)
Extravasation (General disorders) | 1 (1) | 0 (0)
Multi-organ failure (General disorders) | 0 (0) | 1 (1)
Stent malfunction (General disorders) | 0 (0) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1) | 0 (0)
Sudden death (General disorders) | 0 (0) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 7 (8) | 8 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 4 (4) | 3 (3)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Idiopathic thrombocytopenic purpura (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Acute prerenal failure (Renal and urinary disorders) | 2 (2) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 1 (1)
Ureteric obstruction (Renal and urinary disorders) | 1 (1) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal colic (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Ureteric stenosis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Cholestasis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Biliary fistula (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholangitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (1) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 1 (1) | 6 (7)
Anaphylactic shock (Immune system disorders) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3)
Hypertensive emergency (Vascular disorders) | 0 (0) | 1 (2)
Aortic stenosis (Vascular disorders) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 2 (3)
Anastomotic complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiopulmonary failure (Cardiac disorders) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Cerebral atrophy (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Phrenic nerve paralysis (Nervous system disorders) | 1 (1) | 0 (0)
Polyneuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Oncologic complication (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 2 (2)
Disorientation (Psychiatric disorders) | 0 (0) | 1 (1)
Drug dependence (Psychiatric disorders) | 0 (0) | 1 (1)
Volume blood decreased (Investigations) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 1 (1) | 0 (0)
Intestinal operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Ureteral stent insertion (Surgical and medical procedures) | 1 (1) | 0 (0)
Epididymitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Chemotherapy (N=409) | Chemotherapy + Bevacizumab (N=401)
Diarrhoea (Gastrointestinal disorders) | 177 (333) | 233 (471)
Nausea (Gastrointestinal disorders) | 170 (294) | 178 (340)
Vomiting (Gastrointestinal disorders) | 104 (162) | 119 (188)
Abdominal pain (Gastrointestinal disorders) | 76 (91) | 89 (126)
Constipation (Gastrointestinal disorders) | 74 (96) | 82 (120)
Stomatitis (Gastrointestinal disorders) | 32 (47) | 40 (69)
Abdominal pain upper (Gastrointestinal disorders) | 22 (31) | 37 (44)
Asthenia (General disorders) | 106 (263) | 106 (246)
Fatigue (General disorders) | 80 (126) | 94 (154)
Mucosal inflammation (General disorders) | 43 (72) | 76 (136)
Pyrexia (General disorders) | 44 (61) | 66 (92)
Oedema peripheral (General disorders) | 26 (30) | 20 (23)
Neutropenia (Blood and lymphatic system disorders) | 86 (159) | 112 (246)
Thrombocytopenia (Blood and lymphatic system disorders) | 51 (102) | 69 (124)
Leukopenia (Blood and lymphatic system disorders) | 35 (62) | 53 (110)
Anaemia (Blood and lymphatic system disorders) | 58 (93) | 41 (58)
Paraesthesia (Nervous system disorders) | 67 (139) | 78 (179)
Neuropathy peripheral (Nervous system disorders) | 52 (99) | 46 (94)
Polyneuropathy (Nervous system disorders) | 43 (67) | 51 (98)
Peripheral sensory neuropathy (Nervous system disorders) | 21 (47) | 32 (58)
Neurotoxicity (Nervous system disorders) | 13 (29) | 27 (53)
Headache (Nervous system disorders) | 15 (20) | 29 (40)
Alopecia (Skin and subcutaneous tissue disorders) | 68 (85) | 71 (92)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 36 (68) | 50 (96)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 (21) | 70 (88)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 (48) | 36 (40)
Cough (Respiratory, thoracic and mediastinal disorders) | 31 (35) | 35 (42)
Decreased appetite (Metabolism and nutrition disorders) | 77 (99) | 79 (105)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (32) | 26 (34)
Nasopharyngitis (Infections and infestations) | 18 (20) | 28 (33)
Urinary tract infection (Infections and infestations) | 21 (28) | 21 (24)
Hypertension (Vascular disorders) | 24 (29) | 47 (72)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (29) | 30 (39)
Weight decreased (Investigations) | 24 (26) | 37 (38)

LIMITATIONS AND CAVEATS:
Patients in the study who were randomized to receive bevacizumab could continue to receive bevacizumab following discontinuation of chemotherapy, thereby minimizing any potential bias introduced by differential follow-up time in the treatment arms.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.